CLINICAL TRIAL: NCT00984503
Title: A Single-site, Randomised, Double-blind, Phase II Trial to Investigate the Safety, Toleration, Systemic Exposure, Accelerated Healing and Anti-scarring Potential of Juvista in Split Skin Graft Donor Sites in Male Subjects Aged 18-85 Years
Brief Title: Investigation of the Accelerated Healing and Anti-scarring Potential of Avotermin (Juvista) in Split Skin Graft Donor Sites
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: John Hutchison, Medical Director, Renovo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN1001-319-1007
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Cicatrix; Wound Healing
Keywords: Cicatrix; Scar; Wound healing; Avotermin; TGF beta 3; Juvista; RN1001
MeSH Terms: conditions — Cicatrix | interventions — TGFB3 protein, human; Transforming Growth Factor beta3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intradermal Juvista (Experimental)
  Interventions: Drug: Avotermin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Intradermal and topical Juvista (Experimental)
  Interventions: Drug: Avotermin
- Intradermal and topical placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avotermin — Intradermal Juvista at 50ng/100μl/cm2 of SSG donor sites (3cm2) once just prior to wounding
  Other Names: Juvista; TGF beta 3; RN1001
  Arms: Intradermal Juvista
Drug: Placebo — Intradermal injection of Placebo at 100μl/cm2 of SSG donor site (3cm2) once just prior to wounding
  Arms: Placebo
Drug: Avotermin — Intradermal Juvista at 50ng/100μl/cm2 of SSG donor site once just prior to wounding, followed by topical Juvista at 100ng/200μl/cm2 after wounding and again at Day 1
  Other Names: Juvista; TGF beta 3; RN1001
  Arms: Intradermal and topical Juvista
Drug: Placebo — Intradermal placebo at 100μl/cm2 of SSG donor site once just prior to wounding, followed by topical placebo at 200μl/cm2 after wounding and again at Day 1
  Arms: Intradermal and topical placebo

SUMMARY:
The purpose of this study is to investigate the accelerated-healing potential of injection or injection plus topical application of Juvista to minor split skin grafts (SSG).

DETAILED DESCRIPTION:
Subjects were allocated into three groups (Group 1, Group 2 and Group 3) with all subjects receiving two 3cm2 SSG donor sites, one to each side of the lower back. Before wounding on Day 0, each site was randomised to receive either an intradermal injection of Juvista (50ng/100μl/cm2), an intradermal injection of Placebo (100μl/cm2) or no injection (Standard Care). After wounding, subjects allocated to Group 2 and Group 3 also received topical Juvista (100ng/200μl/cm2), topical Placebo (200μl/cm2) or Standard Care (Tegaderm dressing only). Topical Juvista and Placebo were held within a Granuflex ring dressing and sealed with a sterile Tegaderm dressing.

On Day 1, subjects in Group 2 and Group 3 received a further topical application of Juvista, Placebo or Standard Care according to the same treatment randomisation as Day 0.

Punch biopsy samples of healing SSG donor sites were harvested from Group 3 subjects on Day 3, 5, 7 or 10, and preserved for histological analysis.

The final study visit for Group 3 subjects was the day of the biopsy visit. Subjects in Group 1 and Group 2 underwent scar assessments at the first follow-up at Month 1 and at Months 2, 3, 4, 5, 6, 9 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy, male subjects aged 18-85 years
* Weight between 40 and 150kg or a BMI within the permitted range for their height using Quetelet's index, 15-55 kg/m2. Weight (kg)/height (m)2.

Exclusion Criteria:

* Subjects who had a history or evidence of hypertrophic or keloid scarring or had tattoos or previous scars in the area of the prospective SSG donor sites
* Subjects who had received surgery to the area of the lower back/buttocks in the previous 12 months
* Afro-Caribbean subjects were excluded because of their increased susceptibility to hypertrophic and keloid scarring
* Subjects who had evidence of any past or present clinically significant disease, particularly coagulation disorders, diabetes, immunomediated conditions, skin diseases and allergies (such as clinically significant eczema
* Subjects with a history of clinically significant allergies, especially drug hypersensitivity to lignocaine, allergy to surgical dressings used in this trial or to any excipients or vehicle in the formulation or delivery vehicle
* Subjects with any clinically significant abnormality following review of pre-trial laboratory data and physical examination
* Subjects who were receiving or had received certain prescribed drugs in the 4 weeks prior to Day 0, particularly topical or systemic steroids, anti- inflammatory, anti-coagulants, antiproliferative drugs and antibiotics. Certain drugs not excluded in this trial included over-the-counter analgesics, including paracetamol and codeine, vitamin and mineral supplements, and cold remedies. If antibiotics were required after Day 0 (e.g., for cases of wound infection), this did not result in the exclusion of affected subjects from the study
* Subjects who had taken part in a clinical trial within 3 months prior to admission to this trial or who are currently participating in a clinical trial, whether an investigational drug was used or not.
* Subjects who had any clinical evidence of severe ongoing or prolonged depression or mental illness
* Subjects who smoked more than 20 cigarettes a day
* Subjects who drank more than 28 units of alcohol per week (1 unit = ½ pint of beer [285ml], 25ml of spirits or 1 glass of wine)
* Subjects who demonstrated evidence of drug abuse
* Subjects who were known to have or have had serum hepatitis and those who are carriers of the hepatitis B surface antigen or hepatitis C antibody (Subjects with previous vaccination against hepatitis B were not excluded per se)
* Subjects who were known to have, or have had, serum hepatitis and those who were carriers of the hepatitis B core antibody with less than 10 units per litre of anti-hepatitis B (unless deemed NOT to be a carrier of hepatitis B after testing by the Public Health Laboratory)
* Subjects who had previously tested positive for HIV antibodies or who admitted to belonging to a high-risk group
* A subject who, in the opinion of the Investigator, was unlikely to complete the trial for whatever reason

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-10; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To assess the accelerated-healing potential of injection or injection plus topical application of Juvista in a male population undergoing minor split skin grafts (SSG) | Up to 12 months

SECONDARY OUTCOMES:
To assess the local safety and toleration of injection of Juvista or injection and topical application of Juvista at the SSG donor site in a healthy male population | Up to 12 months
To assess systemic exposure following injection of Juvista or injection plus topical application of Juvista after SSG | Up to 12 months
To assess the anti-scarring potential of injection or injection and topical application of Juvista in a male population | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Duncan, Principal Investigator — Renovo; Jeremy Bond, Principal Investigator — Renovo; James Bush, Principal Investigator — Renovo
Locations (1):
- Renovo, Manchester, United Kingdom